CLINICAL TRIAL: NCT00240058
Title: Pilot Study On The Role Of Nitric Oxide In Alpha 1-Adrenergic Vasoreactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Crystal A. Gadegbeku (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Michigan (Other)
Responsible Party: Sponsor-Investigator, Crystal A. Gadegbeku, Assistant Professor of Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DRDA05-0222; R33DK071222 (NIH)
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Blood Pressure
Keywords: Blood Pressure; Nitric Oxide; L-NMMA; Phenylephrine; Nitroprusside; Vasoreactivity

ARMS (1):
- phenylephrine infusion with and without nitric oxide clamp (Other): Participants received phenylephrine infusion with saline followed by phenylephrine infusion with nitric oxide clamp
  Interventions: Drug: Regional phenylephrine arterial infusion, Nitric Oxide Clamp

INTERVENTIONS:
Drug: Regional phenylephrine arterial infusion, Nitric Oxide Clamp

SUMMARY:
This is a research project to test two study techniques among healthy adults. The procedures look at how blood flow is controlled by substances in blood vessels.

DETAILED DESCRIPTION:
Most patients with chronic kidney disease (CKD) have high blood pressure and are at high risk for cardiovascular disease. High blood pressure can be partly caused by narrowing of blood vessels from high activity of the alpha1-adrenoceptor system in blood vessels. On the other hand, nitric oxide (NO), produced by the body, opposes the alpha 1-adrenoceptor system. NO widens blood vessels and prevents high blood pressure. We hypothesize that low availability of NO may be responsible for high activity of alpha 1-adrenoceptor system in patients with CKD. This protocol is a pilot study in healthy subjects to guide us in performing future studies in patients with CKD.

The specific aims of the pilot study, in healthy people, are to 1) determine whether alpha 1-adrenoceptor vasoreactivity is reproducible and 2) determine alpha 1-adrenoceptor vasoreactivity with the NO clamp technique. To carry out these specific aims, we will consent and enroll healthy people with normal blood pressure. After a screening visit to confirm eligibility, subjects will be admitted to the General Clinical Research Center overnight for a study the following day.

We will constrict the forearm blood vessels by giving different amounts of phenylephrine into the artery through a catheter. We will measure the subjects blood flow with venus plethysmography ( a measuring tool like a blood pressure cuff) while giving the phenylephrine. We will repeat the tests to see if we get the same results.

Then, a research medication, L-NMMA, which blocks NO in the blood vessel, will be dripped into the same artery followed by another medication nitroprusside, which gives back NO, to restore normal forearm blood flow. This procedure is called the NO clamp technique and is used to measure the effects of NO. The phenylephrine concentrations and plethysmography will be repeated again to compare vessel narrowing before and during the NO clamp. This research will teach us how to perform future studies on the relationship between NO and the alpha 1-adrenoceptor system in patients with kidney disease.

ELIGIBILITY:
Inclusion Criteria:

Healthy men and women:

* Age 18 to 55 years
* Who have Blood Pressure less than or equal to 120/80.

Exclusion Criteria:

Individuals with:

* Diabetes, lung disease
* Stomach disease, liver disease
* Blood vessel disease
* Kidney disease
* High blood pressure
* Heart disease
* Hereditary blood disorders
* Hematocrit (amount of red blood cells) less than 30%,
* Who smoke
* Women who are pregnant or lactating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2005-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Determine whether alpha 1-adrenoceptor vasoreactivity is reproducible
Determine alpha 1-adrenoceptor vasoreactivity with the NO clamp technique

CONTACTS AND LOCATIONS:
Overall Officials: Crystal A Gadegbeku, MD, Principal Investigator — Assistant Professor of Medicine, University of Michigan Health System, Department of Internal Medicine, Division of Nephrology
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- See also: Principle Investigator research information — http://www.med.umich.edu/intmed/nephrology/STAFF/gadegbeku_ca1.htm